CLINICAL TRIAL: NCT00599066
Title: Same-patient Reproducibility of Intraoperative M-Entropy Measurements
Brief Title: Intraoperative M-Entropy Measurements
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: IRB No: 13577
Record Dates: First submitted 2007-12-20; First posted 2008-01-23 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: General Anesthesia
Keywords: M-Entropy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study cases: Application of a second M-Entropy probe on the forehead of the patient; at the end the patient will have 2 probes on the forehead, one in the right and one in the left.
  Interventions: Device: study cases

INTERVENTIONS:
Device: study cases — Application of a second M-Entropy probe on the forehead of the patient, which will happen in the OR along with the application of other monitors immediately before induction of general anesthesia.
  Other Names: M-entropy module (Datex-Ohmeda S/5 EntropyTM Module)

SUMMARY:
The purpose of this study is to learn more about an Entropy monitor that the anesthesiologist will be using.

DETAILED DESCRIPTION:
Depth of anesthesia monitors are increasingly used in clinical anesthesia practice. Bispectral Index (BIS) and M-Entropy are examples to these devices, both of which are available at our institution. Both BIS and M-Entropy use a unilateral, single channel of EEG to derive a number indicating the anesthetic depth. These devices have similar disposable skin probes that can be applied on either side of the forehead. Since the depth of anesthesia for an individual is the same over the whole brain cortex at a given point in time, BIS numbers obtained over the left and right side of the forehead should agree. The same should be true for M-Entropy as well.

A recent study, however, showed that two separate BIS probes, applied over the left and right forehead of the same patient at the same time, can give significantly different numbers. This has not been studied for M-Entropy. BIS and M-Entropy use different mathematical algorithms that process the raw EEG signal to compute a numeric value. Therefore, it is possible that M-Entropy may show different results in a similar study setup.

The aim is to investigate the same-patient reproducibility of M-Entropy by monitoring and recording Entropy variables over both the left and the right side of the forehead of patients under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to have surgery under general anesthesia, with a minimum of 60 minutes expected duration.

Exclusion Criteria:

* Non-English speaker
* Patients younger than 18 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are scheduled to have surgery under general anesthesia for which an intraoperative M-Entropy monitoring is planned. Suitable candidates will be identified by speaking to the attending anesthesiologists working at OU Presbyterian hospital.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The investigators hypothesize that simultaneous M-Entropy measurements from the left and right side of the forehead of a person do not differ during general anesthesia. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mehemet Ozcan, MD, Principal Investigator — The University of Oklahoma Health Sciences Center, Department of Anesthesiology
Locations (1):
- OU MEDICAL CENTER, Presbyterian Tower, OR, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niedhart DJ, Kaiser HA, Jacobsohn E, Hantler CB, Evers AS, Avidan MS. Intrapatient reproducibility of the BISxp monitor. Anesthesiology. 2006 Feb;104(2):242-8. doi: 10.1097/00000542-200602000-00007. PMID 16436841
- [Background] Ozcan MS, Gravenstein D. The presence of working memory without explicit recall in a critically ill patient. Anesth Analg. 2004 Feb;98(2):469-470. doi: 10.1213/01.ANE.0000096184.32247.D0. PMID 14742389